CLINICAL TRIAL: NCT02974205
Title: Kneelaxity and Self-reported Knee Function After Rehabilitation With the Use of Dynamic Kneeorthosis for Patients With Acute Isolated Posterior Cruciate Ligament Injury: A Randomized Controlled Trial
Brief Title: Rehabilitation of Patient With Acute Isolated PCL Rupture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Ingrid Trøan, PT, MSc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 579239
Record Dates: First submitted 2016-11-17; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: PCL
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rehabilitation with orthosis (Jack brace) (Active Comparator)
  Interventions: Procedure: Jack brace
- Rehabilitation without orthosis (Active Comparator)
  Interventions: Device: Rehabilitation
- Rehabilitation with orthosis (össur brace) (Active Comparator)
  Interventions: Device: össur brace

INTERVENTIONS:
Procedure: Jack brace — Rehabilitation after acute isolated PCL rupture with orthosis
  Arms: Rehabilitation with orthosis (Jack brace)
Device: Rehabilitation — Rehabilitation after acute isolated PCL rupture without orthosis
  Arms: Rehabilitation without orthosis
Device: össur brace — Rehabilitation after acute isolated PCL rupture
  Arms: Rehabilitation with orthosis (össur brace)

SUMMARY:
The posterior cruciate ligament injuries (PCL) is rare and rehabilitation methods are varying. The purpose of the study is to explore if one rehabilitation option is preferable to one other for patients with acute PCL injury, by examining whether there will be differences in laxity in the knee joints and patient-reported knee function by three different rehabilitation protocols. A randomized controlled trial with 75 patients enrolled will be followed up 3 and 12 months after injury. The groups will be compared using kneelaxity (stress - X) and subjective knee function (KOOS, IKDC-2000)

DETAILED DESCRIPTION:
The posterior cruciate ligament injuries (PCL) is rare and rehabilitation methods are varying. The purpose of the study is to explore if one rehabilitation option is preferable to one other for patients with acute PCL injury, by examining whether there will be differences in laxity in the knee joints and patient-reported knee function by three different rehabilitation protocols. A randomized controlled trial with 75 patients enrolled will be followed up 3 and 12 months after injury. The groups will be compared using kneelaxity (stress - X) and subjective knee function (KOOS, IKDC-2000) to indicate whether one rehabilitation alternative is preferable in terms of less knee joint laxity and improve knee function. Participants considered included in the study if he or she agrees to participate in the study by signing the informed consent. Inclusion criteria will be whether the patient has an acute isolated PCL injury. Exclusion is additional injuries of ligaments, cartilage and meniscus of the knee. Randomization to groups is done continuously.

ELIGIBILITY:
Inclusion Criteria:

* Acute isolated PCL injury : 0- 3 weeks ( maximum 21 days) from the initial injury
* Isolated PCL rupture (grade I, II and III)
* Patient age should be between 16-60 years ( with closed epiphyseal plate )
* Understood and accepted written consent

Exclusion Criteria:

* Injury to the ACL or other ligaments in the knee
* Extensive injury to the cartilage or meniscus , requiring repairs
* Unfit to understand or to sign consent
* History of alcohol or drug abuse in the past three years
* Current serious illness or injury that makes rehabilitation difficult.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
PCL stress-radiograph | 12 month

SECONDARY OUTCOMES:
KOOS (Knee Injury and Osteoarthritis Outcome score) | 12 month
IKDC-2000 (Subjective Knee Evaluation Form) | 12 month
One leg hop (in meters) | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Lars Engebretsen, Dr. Med, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No